CLINICAL TRIAL: NCT03596632
Title: A Phase 1 Open-label Study Investigating the Excretion Balance, Pharmacokinetics, and Metabolism of a Single Oral Dose of [14C/12C]-Labeled Fenebrutinib in Healthy Volunteers
Brief Title: Study Investigating a Single Oral Dose of Fenebrutinib in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GP40605
Record Dates: First submitted 2018-07-13; First posted 2018-07-24 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2018-12

CONDITIONS: Healthy Participants
MeSH Terms: interventions — fenebrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Oral Solution Dose (Experimental): Single 200-mg (approximately 100-µCi) oral solution dose of [14C/12C]-fenebrutinib under fasted conditions.
  Interventions: Drug: Fenebrutinib

INTERVENTIONS:
Drug: Fenebrutinib — 200-mg (100 µCi) oral solution 14C/12C]-fenebrutinib
  Other Names: RO7010939

SUMMARY:
The purpose of this study is to determine the excretion kinetics and mass balance of fenebrutinib in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects, between 18 and 60 years of age, inclusive
* Within body mass index range 18 to 32 kg/m2, inclusive
* In good health, determined by no clinically significant findings from medical history, 12-lead electrocardiogram (ECG), vital signs, and physical examination
* For males who are sterile: agreement to use a condom with a fertile or pregnant female partner from Day -1 until 90 days following Study Completion; for males who are fertile: agreement to use a condom with spermicide with a fertile or pregnant female partner from Day -1 until 90 days following Study Completion

Exclusion Criteria:

* History or symptoms of any significant disease
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator
* History of stomach or intestinal surgery or resection, except appendectomy, hernia repair, and cholecystectomy
* History of malignancy, except for non-melanoma skin carcinoma with 3-year disease-free follow-up
* Participation in any other investigational study drug trial in which receipt of an investigational study drug occurred within 30 days or 5 half-lives, whichever is longer, prior to Day -1
* Exposure to significant diagnostic or therapeutic radiation or current employment in a job requiring radiation exposure monitoring within 12 months prior to Day -1
* Participation in a radiolabeled drug study in which exposures are known to the Investigator within 4 months prior to Day -1, or participation in a radiolabeled drug study in which exposures are not known to the Investigator within 6 months prior to Day -1. The total 12-month exposure from this study and a maximum of 2 other studies must be within the Code of Federal Regulations (CFR) recommended levels considered state (per 21 CFR 361.1), e.g. less than 5,000 mrem whole body annual exposure

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 8 (Actual)
Dates: Start 2018-07-27 (Actual); Primary Completion 2018-08-23 (Actual); Study Completion 2018-08-23 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) Percentage of the Total Radioactive Dose Administered Excreted from Urine and Feces"; TimeFrame: "Day 1 to end of study (approximately 35 days post-dose) | Screening to end of study (approximately 35 days post-dose)
  An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A SAE is defined as any AE that can be fatal, life threatening, prolongs inpatient hospitalization, significant disability, congenital anamoly, is a significant medical event in the Investigator's judgment.

SECONDARY OUTCOMES:
Maximum Observed Concentration (Cmax) of Fenebrutinib and its Metabolites | Day 1 pre-dose to end of study (approximately 35 days post-dose)
Time to Observed Maximum Concentration (Tmax) of Fenebrutinib and its Metabolites | Day 1 pre-dose to end of study (approximately 35 days post-dose)
Area Under the Concentration-Time Curve From Hour 0 to the Last Measurable Concentration (AUC0-t) of Fenebrutinib and its Metabolites | Day 1 pre-dose to end of study (approximately 35 days post-dose)
Area under the Concentration-Time Curve Extrapolated to Infinity (AUC0-infinity) of Fenebrutinib and its Metabolites | Day 1 pre-dose to end of study (approximately 35 days post-dose)
Cumulative Percent of Total Radioactivity Excreted in Urine Over the Sampling Interval (Total % Feu) | Day 1 pre-dose to end of study (approximately 35 days post-dose)
Cumulative Percent of Total Radioactivity Excreted in Feces Over the Sampling Interval (Total % Fef) | Day 1 pre-dose to end of study (approximately 35 days post-dose)
Number of Participants With Clinical Significant Changes in Vital Signs | Screening up to Day 31
  Vital signs incudes oral temperature, respiratory rate, supine blood pressure and pulse.
Number of Participants With Clinical Significant Changes in Physical Examination Findings | Day -1, 28
  Physical examination will consist of an assessment of general appearance, skin, thorax/lungs, abdomen, lymph nodes, head, ears, eyes, nose, throat, neck (including thyroid); and cardiovascular, musculoskeletal, and neurological systems.
Number of Participants With Clinical Significant Changes in Clinical Laboratory Results | Screnning, Day -1, 2, 4, 28
  Laboratory analysis include chemistry panel, complete blood count and urinalysis.
Number of Participants With Clinical Significant Changes in Electrocardiograms (ECGs) | Screening, Day-1, 1 (Pre-dose; 1, 3 hours [h] post-dose), 28, 31

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Covance Clinical Research Unit, Inc, Madison, Wisconsin, United States